CLINICAL TRIAL: NCT04310215
Title: A Multi-center, Single-blind, Randomized, Phase III Clinical Trial to Evaluate the Efficacy and Safety of Adding CARTISTEM® on Microfracture in Patients With Talar Chondral or Osteochondral Defect
Brief Title: Efficacy and Safety of Allogenic Stem Cell Product(CARTISTEM®) for Osteochondral Lesion of Talus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hyundai Bioland Co., Ltd. (Industry)
Collaborators: Medipost Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CARTISTEM_2019_01
Record Dates: First submitted 2020-03-12; First posted 2020-03-17 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-08

CONDITIONS: Chondral or Osteochondral Lesion of Talus
Keywords: OLT; Talus; Chondral Lesion; Osteochondral Lesion; Human umbilical cord blood-derived stem cell; MSC; Mesenchymal stem cell
MeSH Terms: interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Intervention Model Description: A multicenter, Single-blinded, Stratified randomized
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microfracture + CARTISTEM® (Experimental): CARTISTEM® is added on the lesion as a single dose of 500 ㎕/㎠ according to the defect size after arthroscopic curettage and microfracture.
  Interventions: Biological: CARTISTEM®
- Microfracture (Active Comparator): Standard treatment of arthroscopic curettage and microfracture is performed for cartilage defect.
  Interventions: Procedure: Microfracture

INTERVENTIONS:
Biological: CARTISTEM® — *Stratified randomization by lesion size below 1.5㎠ or more than 1.5㎠
  1. Procedure: Microfracture
  2. Biological: CARTISTEM®(Human Umbilical Cord Blood-derived Mesenchymal Stem Cell product)
  Arms: Microfracture + CARTISTEM®
Procedure: Microfracture — *Stratified randomization by lesion size below 1.5㎠ or more than 1.5㎠
  1. Procedure: Microfracture
  Arms: Microfracture

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of adding CARTISTEM®(allogenic umbilical cord blood-derived stem cell product) on microfracture, a currently standard treatment for OLT, in patients with talar chondral or osteochondral defect.

ELIGIBILITY:
Inclusion Criteria:

1. Talar chondral/osteochondral lesion confirmed by radiographical exam at screening or diagnosis, an AOFAS score of 75 or below
2. Ankle joint pain/stiffness with no response to conservative treatment for more than 12 weeks
3. Ankle joint cartilage injury of defect of ICRS grade Ⅳ in MRI
4. Male or female aged more than 18
5. A one-sided lesion
6. Appropriate function of blood clot: PT(INR) < 1.5×ULN, aPTT <1.5×ULN
7. Appropriate renal function: Creatinine ≤ 2.0 ㎎/㎗, Proteinuria ≤ trace
8. Appropriate hepatic function: Total bilirubin ≤ 2.0 ㎎/㎗, AST/ALT ≤ 100 IU/L
9. No evidence of auto-immune disorder: According to investigator's judgement based on relevent symtom and physical exam, anti-nuclear antibody and anti-thyroglobulin antibody tests are able to performed and confirmed negative (If positive, there are possible cases according to diagnostic opinion of medical department)
10. No surgery or radiotherapy for the same ankle joint within 6 weeks
11. Female patients agreeing with maintenance of contraception* during study period

    *hormone contraceptive, implants of intrauterine device or intrauterine system, double barrier contraception[Concurrent use of diaphragm or cervical occlusive cap and male condom], surgical sterilisation, etc.
12. No chronic ligament instability more than grade Ⅲ (Grade 0: none, Grade Ⅰ: 1~5㎜, GradeⅡ: 5~10㎜, Grade Ⅲ: >10㎜)
13. Patients agreeing with participation in this study and signed on informed consent by their own will

Exclusion Criteria:

1. Degenerative arthritis in ankle(Kellgren Lawrence Grade 3-4)
2. Autoimmune disease
3. Infectious disease need to administration of parenteral antibiotics
4. Myocardial infarction, congestive heart failure, other serious cardiac disorder or uncontrolled resistant hypertension
5. Serious medical disease(Ex. Kidney disease such as chronic renal failure or Glomerulonephritis, etc., acute/chronic liver disease such as liver cirrhosis, fatty liver etc., medical history of malignancy*)

   *Complete remission status is possible.
6. Pregnancy or breast-feeding
7. Psychiatric history or epilepsy
8. Alcohol abuse
9. Heavy smoker
10. Chronic inflammatory disease such as rheumatoid arthritis
11. Participants other clinical trials within 4 weeks
12. Administration of immunosuppressing agents such as Cyclosporin A or azathioprine within 6 weeks
13. Patients with acute ligament injury and clinically significant chronic ligament instability
14. Patients treated with surgery or cell therapy product for the same disease
15. Patients with hypersensitivity or allergy history to bovine protein, hyaluronic acid and gentamicin
16. Other inappropriate patients determined by the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
ICRS-Cartilage Repair Assessment Total Score | Week 48
  Arthroscopic evaluation of articular cartilage repair
  : The score range from 12(normal) to 1(severely abnormal) where lower scores indicate more severity of injury

SECONDARY OUTCOMES:
ICRS-Cartilage Repair Assessment Overall Grade | Week 48
  The grades range from 1(normal) to 4 (severely abnormal) where lower grades indicate more complete repair
Improvement degree of Cartilage Repair by MRI | Week 0 and 48
  Changes in MOCART(Magnetic resonance Observation of Cartilage Repair Tissue) score
  : MOCART score is a 9-part and 29-item scoring system, also resulting in a find cartilage repair tissue score between 0 and 100 points. 100 points represent the best imaginable score
Degree of Functional improvement in FAOS(Foot & Ankle Outcome Score) | Week 0, 24 and 48
  : FAOS consists in 42 items that cover 5 dimensions (symptoms, pain, activities of daily living, sport and recreation activities, and quality of life. Raw scores of each sub-scales results of the sum of each items. A normalized score (100 indicationg no symptoms and 0 indicating extreame sysmptoms) is calculated for each subscale
Degree of Functional improvement in AOFAS(The American Orthopaedic Foot & Ankle Score) | Week 0, 24 and 48
  : AOFAS consists in 9 items that can be divided into 3 sub-scales (pain, function and alignment). 100 points of 1 to 100 represent no symptoms or impairments
Degree of Functional improvement in Tegner activity score | Week 0, 24 and 48
  : Tegner activity represents the highest level of activity on scale of 0 to 10 that you are able to participate in currently . The higher values represent a better outcome
Degree of Quality of Life improvement in SF-36(Short Form Health Survey-36) | Week 0, 24 and 48
  : SF-36 comprises 36 items divided into two components of physical health and mental health. Higher scores between 0 and 100 represent better health status
Degree of pain improvement in 100 mm VAS(Visual Analogue Scale) | Week 0, 24 and 48
  * VAS represents higher scores mean higher pain
  * 0 mm (no pain) and 100 mm (worst pain)

CONTACTS AND LOCATIONS:
Locations (6):
- South Korea (6):
  - Kyunghee University Medical Center, Seoul, Dongdaemun-gu
  - Gangnam Severance Hospital, Seoul, Gangnam-gu
  - Samsung Medical Center, Seoul, Gangnam-gu
  - Korea University Guro Hospital, Seoul, Guro-gu
  - Chungnam National University Hospital, Daejeon, Jung-gu
  - Inha University Hospital, Incheon, Jung-gu

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to other researchers.